CLINICAL TRIAL: NCT04899180
Title: Prevalence of Transthyretin Cardiac Amyloidosis in Clinically Significant Aortic Stenosis: A Community Study
Brief Title: Prevalence of Transthyretin Cardiac Amyloidosis in Clinically Significant Aortic Stenosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Omar Abou Ezzeddine, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-004778
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Aortic Stenosis; Transthyretin Amyloidosis; Transthyretin Amyloid Cardiomyopathy; Transthyretin Cardiac Amyloidosis
MeSH Terms: conditions — Aortic Valve Stenosis; Amyloidosis, Hereditary, Transthyretin-Related | interventions — Technetium Tc 99m Pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPECT/CT (Other): 99mTc-PYP single-photon positive emission computed tomography with computed tomography
  Interventions: Drug: 99mTc-PYP

INTERVENTIONS:
Drug: 99mTc-PYP — Radioisotope used by SPECT/CT imaging

SUMMARY:
The purpose of this study is to determine the prevalence of transthyretin cardiac amyloidosis (TTR-CA) among patients with moderate and severe aortic stenosis in Southeast Minnesota using 99mTc-PYP single-photon positive emission computed tomography with computed tomography (SPECT/CT).

DETAILED DESCRIPTION:
Residents of Southeast Minnesota over 75 years of age with an inpatient or outpatient diagnosis of moderate or severe aortic stenosis will be consecutively identified using an automated bi-weekly review of the echo lab calendar (on Mondays and Fridays) at Mayo Clinic Rochester (MCR) and Mayo Clinic Health System (MCHS) sites. Participants will be consented to undergo venipuncture, urine collection and 99mTc-PYP SPECT/CT imaging to rule in/out the diagnosis of TTR-CA. Hence, the prevalence of TTR-CA will be defined. To place this prevalence in perspective of the global aortic stenosis cohort in the community, a rigorous screening log will be maintained to allow generation of a comprehensive CONSORT diagram. Importantly, baseline characteristics of patients who qualify for our study but decline to consent will still be collected provided that consent for use of their records for medical research had previously been granted.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Southeastern Minnesota (Olmsted, Dodge, Fillmore, Mower, Freeborn, Wabasha, or Steele County)
* Age ≥ 75 years
* Current diagnosis of moderate or severe aortic stenosis by most recent (within 6 months at most) echocardiogram as defined by:

  * Moderate AS: 1.0 cm2 < aortic valve area (AVA) ≤ 1.5 cm2
  * Severe AS: AVA ≤ 1.0 cm2

Exclusion Criteria:

* Any cardiac surgery or major chest trauma within 4 weeks of PYP scan
* Myocardial infarction within 4 weeks of PYP scan defined by typical angina, EKG changes and significant change in serial troponins. (Note that chronic troponin elevation is extremely common in cardiac amyloidosis).
* Prior or current exposure to Plaquenil (Hydroxychloroquine)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of TTR-CA in patients with moderate and severe aortic stenosis | Baseline
  Determine the prevalence of Transthyretin Cardiac Amyloidosis in a community based cohort of consecutive patients with moderate or severe aortic stenosis using 99mTc-Pyrophosphate (99mTc-PYP) single-photon positive emission computed tomography with computed tomography (SPECT/CT)

CONTACTS AND LOCATIONS:
Overall Officials: Omar F Abou Ezzeddine, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials